CLINICAL TRIAL: NCT01878474
Title: A Randomised, Double-blind, Placebo-controlled, First Time-in-humans Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single, Escalating Doses of TA-8995 in Healthy Subjects
Brief Title: Evaluation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TA-8995 With Single, Escalating Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TA-8995-01
Record Dates: First submitted 2013-06-04; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Dyslipidemia
Keywords: MT-8995; Dyslipidemia; Cholesteryl ester transfer proteins
MeSH Terms: conditions — Dyslipidemias | interventions — TA-8995

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Single ascending dose in Caucasian men (Experimental)
  Interventions: Drug: TA-8995
- Age-effect in Caucasian men (Experimental)
  Interventions: Drug: TA-8995
- Gender-effect in Caucasian women (Experimental)
  Interventions: Drug: TA-8995
- Single ascending dose in Japanese men (Experimental)
  Interventions: Drug: TA-8995
- Placebo: Single ascending dose in Caucasian men (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo: Age-effect in Caucasian men (Placebo Comparator)
  Interventions: Drug: Placebo
- Placeo: Gender-effect in Caucasian women (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo: Single ascending dose in Japanese men (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TA-8995 — TA-8905 5, 10, 25, 50 (fasted and fed), 100 and 150 mg
  Arms: Single ascending dose in Caucasian men
Drug: TA-8995 — Drug: TA-8995 25 mg
  Arms: Age-effect in Caucasian men
Drug: TA-8995 — Drug: TA-8995 25 mg
  Arms: Gender-effect in Caucasian women
Drug: TA-8995 — Drug: TA-8995 25, 50, 100 and 150 mg
  Arms: Single ascending dose in Japanese men
Drug: Placebo — Single ascending dose in Caucasian men
  Arms: Placebo: Single ascending dose in Caucasian men
Drug: Placebo — Age-effect in Caucasian men
  Arms: Placebo: Age-effect in Caucasian men
Drug: Placebo — Gender-effect in Caucasian women
  Arms: Placeo: Gender-effect in Caucasian women
Drug: Placebo — Single ascending dose in Japanese men
  Arms: Placebo: Single ascending dose in Japanese men

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single doses of TA-8995 in healthy Caucasian and Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men aged 18-55 years and ≥65 years
* Women of non-childbearing potential
* Japanese men aged 18-55 years
* Subjects were deemed healthy on the basis of medical history, physical examination, Electrocardiogram (ECG), vital signs and safety tests of blood and urine
* Subjects were able to give fully informed written consent

Exclusion Criteria:

* HDL-C level ≥2.59 mmol/L
* Abnormal Holter ECG
* Family history of long QT syndrome, hypokalaemia or Torsade de Pointes
* Vital signs or 12-lead ECG values outside the acceptable range
* Positive tests for hepatitis B and C, HIV 1 and 2
* Positive urine pregnancy test (women only)
* Severe adverse reaction or allergy to any drug
* Drug or alcohol abuse
* Smoking within the 6 months before dosing with TA-8995 (Caucasian subjects), or smoking more than 10 cigarettes daily (Japanese subjects)
* Over-the-counter or prescribed medication up to 7 days or 5 half-lives (whichever was longer) before dosing with TA-8995
* Consuming food or drinks containing grapefruit or cranberry within the 7 days before dosing
* Participation in other clinical trials, or loss of more than 450 mL blood within the previous 3 months
* Clinically relevant abnormal findings at the screening assessment
* Clinically relevant abnormal medical history or concurrent medical condition
* Possibility that volunteer would not cooperate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 336 hours post dose
Laboratory tests (haematology, biochemistry and urinalysis) | 336 hours post dose
Vital signs (supine systolic and diastolic blood pressure, heart rate and body temperature) | 336 hours post dose
Peak concentration (ng/mL) of TA-8995 | 336 hours post dose
Time of peak concentration (hr) of TA-8995 | 336 hours post dose
Area under the concentration-time curve (mg/L・hr) up to 24 h (AUC0-24), 72 h (AUC0-72), 168 h (AUC0-168), 336 h (AUC0-336) and infinity (AUC0-∞) of TA-8995 | 336 hours post dose

SECONDARY OUTCOMES:
Plasma Cholesterol Ester Transfer Protein (CETP) activity (%) and concentration (mg/mL) | 336 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Steve Warrington, MA MD FRCP FFPM, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom